CLINICAL TRIAL: NCT00208689
Title: A Review of the Diagnosis, Treatment and Outcomes of Children With Critical Congenital Heart Defects
Brief Title: Critical Congenital Heart Defect (CHD) Outcomes in Children
Status: Terminated | Type: Observational
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Martha L. Clabby, MD, Principal Investigator, Emory University
Other Study IDs: 1058-2003
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2014-02-13 (Estimated); Status verified 2014-02

CONDITIONS: Congenital Heart Disease
Keywords: pediatric; congenital heart disease
MeSH Terms: conditions — Heart Defects, Congenital

SUMMARY:
Congenital heart disease in infants and children often challenges healthcare providers both in regards to diagnosis and in the management of these conditions. The field becomes more complicated as one examines the myriad of defects that present and the complex care that is required. Over the last 20-25 years, the remarkable advances in the medical and surgical management of the most complex lesions have decreased neonatal mortality, such that many more survive the neonatal period. Therefore, new challenges regarding the continued care of this patient cohort of high-risk infants and children exist. In order to continue the improvement of treatment(s) offered to these patients, continuous review and analysis of the current standard of care is needed.

In this study, the investigators will collect information related to the current surgical and medical therapies offered to patients enrolled in the High Risk Congenital Heart Program at Children's Healthcare of Atlanta. All of the procedure and visit information will be a part of the child's standard of care. This information will be placed in a database. The investigators hope to learn more about the short-term and long-term effects of current therapies and procedures.

DETAILED DESCRIPTION:
Patients, age newborn to 21 years, followed in the High Risk Congenital Heart Defect Clinic at Children's Healthcare of Atlanta at Egleston will be asked to participate in this trial. The term "high risk" is assigned to a patient with the following diagnoses or medical problems: critical aortic stenosis, truncus arteriosus (with or without interrupted aortic arch), patients with complex single ventricle physiology (such as hypoplastic left heart syndrome, unbalanced AV canal, tricuspid atresia, transposition of the great vessels with ventricular septal defect and pulmonary stenosis, mitral atresia, pulmonary atresia with intact ventricular septum), left ventricular outflow tract obstruction requiring Konno procedure, transposition of the great vessels (with or without ventricular septal defect), pulmonary atresia with ventricular septal defect, interrupted aortic arch (with or without ventricular septal defect), anatomy requiring "double switch" procedure, aortic arch abnormality requiring transverse arch graft, total anomalous pulmonary venous return, anatomy requiring any of the following procedures: Damas-Kaye-Stansel procedure, ventricular septal defect enlargement, or resection of subpulmonic stenosis during arterial switch procedure, atrial septectomy, neonatal repositioning of the tricuspid valve for Ebstein anomaly, Ross procedure in infancy; mitral stenosis with mitral valve replacement in infancy, and any other cardiac abnormality requiring surgical repair in infancy with residual hemodynamically significant lesions. In addition, patients with infantile Marfan syndrome, or kawasaki disease with coronary artery aneurysm will also be included.

Informed consent will be obtained from the parent or legally authorized representative for all study participants. An Assent, either verbal or written, will also be obtained if the child is over the age of six (6). A sequential and unique subject number (i.e. NES.001, NES.002) will be assigned by the investigator or designee to each qualified subject after informed consent has been obtained. Once a subject number is assigned, it will not be used again by the investigator. Subjects who are asked to participate but refuse participation in the study will not be assigned a study number.

Investigational Plan:

A single-center, retrospective registry design will be utilized. After consent, the following data will be collected from each study participant's chart each time he or she attends clinic:

* Name
* Contact information (or confirm contact information)
* Names of other care providers
* Primary Diagnosis
* Secondary Diagnoses
* Age at time of visit
* Vital signs including blood pressure, heart rate, respirations, pulse oximetry
* Weight at time of visit
* If applicable, echocardiography data including m-mode, tissue doppler and color flow Doppler
* History and Physical including surgical history
* Medications
* Nutritional Status
* Growth Parameters
* If applicable, most recent standard of care laboratories
* If applicable, MRI results
* EKG findings

All procedures are standard of care. The collection of data for this registry will not effect the care provided to each patient. The individual physician has the right to diagnose and treat each patient according to standard of care procedures and his/her own medical judgement.

Participation in this registry will last as long as the patient is being followed in the high risk clinic at Children's Healthcare of Atlanta.

ELIGIBILITY:
Inclusion Criteria:

* Critical congenital heart disease
* Signed informed consent

Exclusion Criteria:

* Not diagnosed with critical congenital heart disease
* No signed informed consent

Ages: 1 Day to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 150
Dates: Start 2004-01; Primary Completion 2006-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martha Clabby, MD, Principal Investigator — Emory University and Children's Healthcare of Atlanta
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States